CLINICAL TRIAL: NCT03452072
Title: Efficacy and Safety of 0.25% Timolol Gel in Healing Surgical Open Wounds: A Randomized Controlled Trial
Brief Title: Efficacy and Safety of 0.25% Timolol Gel in Healing Surgical Open Wounds
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Chrysalyne D Schmults, MD, MSCE, Director, Mohs and Dermatologic Surgery Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BWHMDSC001
Record Dates: First submitted 2018-02-16; First posted 2018-03-02 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Wound of Skin; Wound Heal; Wound Open; Surgical Wound
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: The protocol will begin post-surgery. Eligible subjects will be assigned by computer-based randomization to case (0.25% timolol gel) or control (standard of care [SOC]) group and treated as follows:
  Case group:
  1. Timolol 0.25% gel will be applied to wound bed immediately after surgery before dressing is applied
  2. Starting the day after surgery: each day, the patient will cleanse the surgical site, apply 0.25% topical timolol gel (1 drop = 0.1ml for each cm2 of wound area), and re-cover wound with clean dressing
  3. Daily routine continues for 12 weeks' post-surgery (even if the surgical defect has completely healed)
  SOC group:
  1. Vaseline will be applied to wound bed immediately after surgery before dressing is applied
  2. Starting the day after surgery: each day, the patient will cleanse the surgical site, apply Vaseline, and re-cover wound with clean dressing
  3. This daily routine continues for 12 weeks' post-surgery (even if the surgical defect has completely healed)
Who Masked: Outcomes Assessor
Masking Description: Blinded physician will assess outcomes from pictures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 0.25% Timolol gel under the paraffin gauzes (Experimental): 1. Timolol 0.25% gel will be applied to wound bed immediately after surgery before dressing is applied
  2. Starting the day after surgery: each day, the patient will cleanse the surgical site, apply 0.25% topical timolol gel (1 drop = 0.1ml for each cm2 of wound area), and re-cover wound with clean dressing
  3. This daily routine continues for 12 weeks' post-surgery (even if the surgical defect has completely healed in the interim)
  Interventions: Drug: 0.25% Timolol gel with paraffin gauze dressings
- Standard of Care dressings (Active Comparator): 1. Vaseline will be applied to wound bed immediately after surgery before dressing is applied
  2. Starting the day after surgery: each day, the patient will cleanse the surgical site, apply Vaseline, and re-cover wound with clean dressing
  3. This daily routine continues for 12 weeks' post-surgery (even if the surgical defect has completely healed in the interim)
  Interventions: Other: Vaseline dressing

INTERVENTIONS:
Drug: 0.25% Timolol gel with paraffin gauze dressings — Timolol 0.25% gel will be applied to wound bed immediately after surgery before dressing is applied. Starting the day after surgery: each day, the patient will cleanse the surgical site, apply 0.25% topical timolol gel (1 drop = 0.1ml for each cm2 of wound area), and re-cover wound with clean dressing
  Arms: 0.25% Timolol gel under the paraffin gauzes
Other: Vaseline dressing — Vaseline will be applied to wound bed immediately after surgery before dressing is applied. Starting the day after surgery: each day, the patient will cleanse the surgical site, apply Vaseline, and re-cover wound with clean dressing
  Arms: Standard of Care dressings

SUMMARY:
The use of topical beta-blockers, such as 0.25% timolol, in promoting wound healing is currently emerging in the academic literature. The investigators will enroll 114 patients who have their skin cancer surgically removed resulting in open surgical wounds less or equal to 1.5 cm. The objective of this randomized safety study is to determine the safety and efficacy of 0.25% timolol in promoting wound healing in open surgical wounds less or equal to 1.5 cm.

DETAILED DESCRIPTION:
Healing of a cutaneous defect by second intention is a complex process. Migration of fibroblasts, keratinocytes, and other cell types to the site of defect and their proliferation under stimulation by cytokines and growth factors occur during this process. The role of topical beta-blockers in promoting wound healing is currently emerging in the international literature (1-3). β2-Adrenergic receptors (B2AR) are the only subtype of beta-adrenoceptors expressed on skin (4-6). They can be found in secretory coil of apocrine glands, keratinocytes, fibroblasts and melanocytes. The distribution of these receptors provides insight on dermatological disorders that may be affected by β-blockers. Keratinocyte migration occurs by the facilitation of chemotaxis, the polarization of cells, and activation of extracellular signal-related kinases essential in the signaling of promigratory pathways. The B2AR activation inhibits keratinocyte migration by activating the serine/threonine phosphatase 2A, which downregulates phosphorylation of extracellular signal-related kinases necessary for migration. Therefore, B2AR antagonists prevent the phosphorylation of phosphatase 2A and have the downstream effect of extracellular signal-related kinase promotion, inducing a promigratory pathway in keratinocytes (4-6). Keratinocyte migration also occurs by galvanotaxis, a phenomenon in which cells migrate in response to electric stimuli. Keratinocytes can be stimulated to migrate with the formation of electrical poles and the application of electrical fields. The B2AR antagonists improve the ability of keratinocytes to respond to such migratory cues, whereas the B2AR agonists decrease keratinocytes' ability to respond, further implicating the use of topical timolol for recalcitrant wounds (4-6). Angiogenesis and dermal fibroblast proliferation are also regulated by B2ARs. The B2AR antagonists have been found to promote angiogenesis in chick chorioallantoic membrane assays and in vivo murine wound models. Dermal fibroblast migration is also increased (by 27%) when exposed to B2AR antagonists, and epidermal differentiation is improved with B2AR antagonists and β1- and β2-receptor antagonists (5-10).

Topical beta-blockers have been gaining increasing popularity and evidence over the last few years as enhancers of wound healing in acute and chronic open wounds. In particular, 0.25% timolol gel may represent a commercially available, safe and simple, painless-though perhaps moderately expensive-treatment for improving both acute and chronic open wounds, as well as for improving long-term cosmetic outcomes.

To assess the efficacy and safety of topically applied 0.25% timolol gel in promoting wound healing in surgical open wounds ≤1.5cm versus standard of care (SOC) by:

1. Evaluating healing in response to treatment with 0.25% topical timolol gel versus SOC in terms of wound surface area reduction of open surgical wound;
2. Evaluating cosmetic outcomes of surgical wounds in terms of blinded physician (Vancouver Scar Scale, VSS) and patient (Visual Analogue Scale, VAS) assessment at 3 and 6 months follow up;
3. Evaluating patient discomfort during the healing process by means of a patient pain VAS;
4. Determining the side effects associated to 0.25% topical timolol versus SOC; and
5. Determining costs associated to the use of 0.25% topical timolol versus SOC.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Open surgical wound ≤1.5cm
3. No hypersensitivity with use of 0.25% timolol gel

Exclusion Criteria:

1. Age less than 18 years of age
2. Open surgical wound >1.5cm
3. Pregnant women
4. Use of systemic retinoids within 1 month
5. Any hypersensitivity with use of 0.25% timolol gel

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in histogram planimetry for open surgical wounds | 7 days' post-surgery, 15 days' post-surgery, 30 days' post-surgery, 3 months' post-surgery, 6 months' post-surgery
  Histogram planimetry is more accessible and less expensive than automated analysis software programs, and it is based on the pixel count of a selected irregular area which is divided by the pixel count of 1 cm2 to find a result in terms of cm2 or mm2

SECONDARY OUTCOMES:
Cosmetic outcomes of open surgical wound healing by blinded physician Vancouver Scar Scale assessment | 3 months' post-surgery, 6 months' post-surgery
  A physician blinded to the treatment group the subject is in will self-administer the Vancouver Scar Scale (VSS) which documents change in scar appearance over time via standardized photographs. The VSS ranges from 0 (most desirable outcome) to 13 (least desirable outcome), thus, a lower score is considered to have a better outcome and a higher score is considered a worse outcome. The VSS consists of four sub-scales, with each sub-scale reporting a value. The "pigmentation sub-scale" ranges from 0 (normal pigmentation) to 2 (hyperpigmentation); the "vascularity sub-scale" ranges from 0 (normal appearance) to 3 (purple appearance); the "pliability sub-scale" ranges from 0 (normal pliability) to 5 (contracture); and the "height sub-scale" ranges from 0 (normal [flat]) to 3 (>5mm). Sub-scale scores are combined to give an overall VSS assessment score.
Study subject complete the Patient Scar Assessment via Visual Analogue Scale | 3 months' post-surgery, 6 months' post-surgery
  Subjects will be asked to complete a Visual Analogue Scale for scar assessment to rate how they think their graft sites appear cosmetically compared to normal skin, and any complaints about how painful they sites are, and how itchy they feel. Each question ranges from 1 (no complaints with itch or pain/as normal skin) to 10 (worst imaginable itch or pain/very different from normal skin). The PSAS ranges from 6 (best outcome score) to 66 (worst outcome score), thus a lower score is considered to have a better outcome and a higher score is considered a worse outcome.
Determine side effects associated with 0.25% topical timolol for open surgical wounds | 7 days' post-surgery, 15 days' post-surgery, 30 days' post-surgery, 3 months' post-surgery, 6 months' post-surgery
  Patients will report and side effects they experience post-surgery. A physician will also assess for side effects and determine whether they are likely associated with the 0.25% topical timolol or part of the normal wound healing experience.

CONTACTS AND LOCATIONS:
Overall Officials: Chrysalyne D Schmults, MD, MSCE, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Mohs and Dermatologic Surgery Center, Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Braun LR, Lamel SA, Richmond NA, Kirsner RS. Topical timolol for recalcitrant wounds. JAMA Dermatol. 2013 Dec;149(12):1400-2. doi: 10.1001/jamadermatol.2013.7135. No abstract available. PMID 24172892
- [Background] Ali A, Herndon DN, Mamachen A, Hasan S, Andersen CR, Grogans RJ, Brewer JL, Lee JO, Heffernan J, Suman OE, Finnerty CC. Propranolol attenuates hemorrhage and accelerates wound healing in severely burned adults. Crit Care. 2015 May 4;19(1):217. doi: 10.1186/s13054-015-0913-x. PMID 25936635
- [Background] Vestita M, Bonamonte D, Filoni A. Topical propranolol for a chronic recalcitrant wound. Dermatol Ther. 2016 May;29(3):148-9. doi: 10.1111/dth.12328. Epub 2016 Jan 22. No abstract available. PMID 26800510
- [Background] Yesiloglu N, Yildiz K, Cem Akpinar A, Gorgulu T, Sirinoglu H, Ozcan A. Histogram Planimetry Method for the Measurement of Irregular Wounds. Wounds. 2016 Sep;28(9):328-333. PMID 27701128
- [Background] Thomas B, Kurien JS, Jose T, Ulahannan SE, Varghese SA. Topical timolol promotes healing of chronic leg ulcer. J Vasc Surg Venous Lymphat Disord. 2017 Nov;5(6):844-850. doi: 10.1016/j.jvsv.2017.04.019. Epub 2017 Aug 7. PMID 29037357
- [Background] Manahan MN, Peters P, Scuderi S, Surjana D, Beardmore GL. Topical timolol for a chronic ulcer--a case with its own control. Med J Aust. 2014 Jan 20;200(1):49-50. doi: 10.5694/mja13.10823. No abstract available. PMID 24438420
- [Background] Lev-Tov H, Dahle S, Moss J, Isseroff RR. Successful treatment of a chronic venous leg ulcer using a topical beta-blocker. J Am Acad Dermatol. 2013 Oct;69(4):e204-5. doi: 10.1016/j.jaad.2013.06.003. No abstract available. PMID 24034405
- [Background] Tang JC, Dosal J, Kirsner RS. Topical timolol for a refractory wound. Dermatol Surg. 2012 Jan;38(1):135-8. doi: 10.1111/j.1524-4725.2011.02200.x. Epub 2011 Oct 31. No abstract available. PMID 22093053
- [Background] Zheng Z, Liu Y, Yang Y, Tang J, Cheng B. Topical 1% propranolol cream promotes cutaneous wound healing in spontaneously diabetic mice. Wound Repair Regen. 2017 May;25(3):389-397. doi: 10.1111/wrr.12546. Epub 2017 May 26. PMID 28494521